CLINICAL TRIAL: NCT02908672
Title: A Phase III, Double-Blinded, Randomized, Placebo-Controlled Study of Atezolizumab Plus Cobimetinib and Vemurafenib Versus Placebo Plus Cobimetinib and Vemurafenib in Previously Untreated BRAFV600 Mutation-Positive Patients With Unresectable Locally Advanced or Metastatic Melanoma
Brief Title: A Study of Atezolizumab Plus Cobimetinib and Vemurafenib Versus Placebo Plus Cobimetinib and Vemurafenib in Previously Untreated BRAFv600 Mutation-Positive Patients With Metastatic or Unresectable Locally Advanced Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CO39262; 2016-002482-54 (EudraCT Number)
Record Dates: First submitted 2016-09-19; First posted 2016-09-21 (Estimated); Results first posted 2020-11-19 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-06

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — atezolizumab; cobimetinib; Vemurafenib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Atezolizumab + Cobimetinib + Vemurafenib + Vemurafenib Placebo (Experimental): Run-In Period (Cycle 1=28 days): Participants will receive vemurafenib 960 mg (four, 240 mg tablets) PO BID along with cobimetinib 60 mg (three, 20 mg tablets) PO QD on Days 1 to 21 followed by vemurafenib 720 mg (three, 240 mg tablets) PO BID on Days 22 to 28 and vemurafenib placebo (1 tablet) PO BID on Days 22 to 28. Triple Combination Period (Cycle 1 onwards): Participants will receive atezolizumab 840 mg IV infusion on Day 1 and 15, cobimetinib 60 mg (three, 20 mg tablets) PO QD on Days 1 to 21, vemurafenib 720 mg (three, 240 mg tablets) PO BID on Days 1 to 28, and vemurafenib placebo (1 tablet) PO BID on Days 1 to 28 of each 28-day cycle. Study treatment will continue until investigator-determined disease progression, death, unacceptable toxicity, withdrawal of consent, or pregnancy, whichever occurs first.
  Interventions: Drug: Atezolizumab; Drug: Cobimetinib; Drug: Vemurafenib; Drug: Vemurafenib Placebo
- Atezolizumab Placebo + Cobimetinib + Vemurafenib (Experimental): Run-In Period (Cycle1=28 days): Participants will receive vemurafenib 960 milligrams (mg) (four, 240 mg tablets) orally (PO) twice a day (BID) along with cobimetinib 60 mg (three, 20 mg tablets) PO once a day (QD) on Days 1 to 21 followed by vemurafenib 960 mg (four, 240 mg tablets) PO BID on Days 22 to 28. Triple Combination Period (Cycle 1 onwards): Participants will receive ATZ placebo by intravenous (IV) infusion on Day 1 and 15, cobimetinib 60 mg (three, 20 mg tablets) PO QD on Days 1 to 21, and vemurafenib 960 mg (four, 240 mg tablets) PO BID on Days 1 to 28 of each 28-day cycle. Study treatment will continue until investigator-determined disease progression, death, unacceptable toxicity, withdrawal of consent, or pregnancy, whichever occurs first.
  Interventions: Drug: Atezolizumab Placebo; Drug: Cobimetinib; Drug: Vemurafenib

INTERVENTIONS:
Drug: Atezolizumab — Will be administered as per the schedule described in individual arm.
  Arms: Atezolizumab + Cobimetinib + Vemurafenib + Vemurafenib Placebo
Drug: Atezolizumab Placebo — Will be administered as per the schedule described in individual arm.
  Arms: Atezolizumab Placebo + Cobimetinib + Vemurafenib
Drug: Cobimetinib — Will be administered as per the schedule described in individual arm.
Drug: Vemurafenib — Will be administered as per the schedule described in individual arm.
Drug: Vemurafenib Placebo — Will be administered as per the schedule described in individual arm.
  Arms: Atezolizumab + Cobimetinib + Vemurafenib + Vemurafenib Placebo

SUMMARY:
This is a Phase III, double-blinded, placebo-controlled, randomized, multicenter study designed to evaluate the efficacy, safety, and pharmacokinetics of atezolizumab + cobimetinib + vemurafenib compared with placebo + cobimetinib + vemurafenib in patients with previously untreated BRAFv600 mutation-positive metastatic or unresectable locally advanced melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Females of child bearing potential and males with female partners must and use of contraceptive methods with a failure rate of less than or equal to (</=)1% per year is required during treatment and for 6 months post treatment. Males should not expose pregnant partners to sperm and refrain from donating sperm for 6 months post treatment. Women must refrain from donating eggs during this same period
* Histologically confirmed Stage IV (metastatic) or unresectable Stage IIIc (locally advanced) melanoma
* Naive to prior systemic anti-cancer therapy for melanoma (example: chemotherapy, hormonal therapy, targeted therapy, immunotherapy, or other biologic therapies) except adjuvant treatment with interferon (IFN), interleukin (IL)-2, or vaccine therapies or herbal therapies
* Documentation of BRAFv600 mutation-positive status in melanoma tumor tissue (archival or newly obtained) through use of a clinical mutation test approved by the local health authority
* Eastern Cooperative Oncology Group Performance (ECOG) Status of 0 or 1
* Measurable disease according to RECIST v1.1 (must be outside central nervous system (CNS))
* Life expectancy >/=18 weeks
* For participants not receiving therapeutic anticoagulation: International normalized ratio (INR) or activated partial thromboplastin time (aPTT) less than or equal to (</=) 1.5*upper limit of normal (ULN) within 28 days prior to initiation of study treatment
* For participants receiving therapeutic anticoagulation: stable anticoagulant regimen and stable INR during the 28 days immediately preceding initiation of study treatment

Exclusion Criteria:

Cancer-Related Exclusion Criteria:

* Major surgical procedure within 4 weeks prior study treatment initiation
* Traumatic injury or palliative radiotherapy within 2 weeks prior study treatment initiation
* Active malignancy (other than BRAFv600 mutation-positive melanoma) or malignancy within 3 years prior to screening are excluded, with the exception of resected melanoma, resected basal cell carcinoma (BCC), resected cutaneous squamous cell carcinoma (SCC), resected carcinoma in situ of the cervix, resected carcinoma in situ of the breast, in situ prostate cancer, limited-stage bladder cancer, or any other curatively treated malignancies from which the participant has been disease-free for at least 3 years

Ocular Exclusion Criteria:

* History of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment, central serous chorioretinopathy, retinal vein occlusion (RVO), or neovascular macular degeneration

Cardiac Exclusion Criteria:

* History of clinically significant cardiac dysfunction
* Left ventricular ejection fraction (LVEF) below the institutional lower limit of normal or below 50%

Central Nervous System (CNS) Exclusion Criteria:

* Untreated or actively progressing CNS lesions (carcinomatous meningitis)
* History of metastases to brain stem, midbrain, pons, or medulla, or within 10 millimeter (mm) of the optic apparatus (optic nerves and chiasm); or leptomeningeal metastatic disease; or intracranial hemorrhage

Additional Exclusion Criteria:

* Uncontrolled diabetes or symptomatic hyperglycemia
* Current severe, uncontrolled systemic disease (including, but not limited to, clinically significant cardiovascular, pulmonary, or renal disease) other than cancer
* History of malabsorption or other clinically significant metabolic dysfunction
* Pregnant or breastfeeding, or intending to become pregnant during the study
* Prior allogeneic stem cell or solid organ transplantation
* History of idiopathic pulmonary fibrosis, organizing pneumonia (example: bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Active or history of autoimmune disease or immune deficiency
* Known clinically significant liver disease, inherited liver disease and active viral disease
* Active tuberculosis
* Treatment with therapeutic oral or intravenous (IV) antibiotics; or with a live, attenuated vaccine; or systemic immunosuppressive medication
* Known hypersensitivity to biopharmaceutical agents produced in Chinese hamster ovary cells or any component of the atezolizumab, cobimetinib, or vemurafenib formulations
* Any grade >/=3 hemorrhage or bleeding event within 4 weeks prior to initiation of study treatment
* History of stroke, reversible ischemic neurological defect, or transient ischemic attack within 6 months prior to initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (110):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Oncology Associates, PC - HAL, Tempe, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - UC Irvine Medical Center, Orange, California
  - Mount Sinai Medical Center, Miami Beach, Florida
  - UF Health Cancer Center at Orlando Health, Orlando, Florida
  - St. Luke's University Health network, Bethlehem, Pennsylvania
- Australia (4):
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (3):
  - Medical University of Graz, Department of Dermatology, Graz
  - LKH Innsbruck, Innsbruck
  - Medizinische Universität Wien, Vienna
- Belgium (4):
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Leuven Gasthuisberg, Leuven
  - CHU Sart-Tilman, Liège
  - Sint Augustinus Wilrijk, Wilrijk
- Brazil (5):
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa e Ensino em Oncologia de Santa Catarina - CEPEN, Florianópolis, Santa Catarina
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Clinicas Oncologicas Integradas - COI, Rio de Janeiro
  - Beneficencia Portuguesa de Sao Paulo, São Paulo
- Canada (8):
  - Arthur J.E. Child Comprehensive Cancer Center-Calgary, Calgary, Alberta
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Juravinski Cancer Clinic, Hamilton, Ontario
  - LHSC - Victoria Hospital, London, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHU de Quebec - Hopital de l'Enfant-Jesus, Québec
- France (7):
  - Groupe Hospitalier Saint André - Hôpital Saint André, Bordeaux
  - Centre Hospitalier Universitaire de Grenoble - Albert Michallon, Grenoble
  - Hopital Claude Huriez - CHU Lille, Lille
  - CHU de Nantes, Nantes
  - Hopital Robert Debre, Reims
  - Centre Eugene Marquis, Rennes
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen
- Germany (18):
  - Charite - Universitätsmedizin Berlin, Berlin
  - Elbekliniken Buxtehude, Buxtehude
  - Klinikum d.Universität zu Köln Klinik u.Poliklinik f.Dermatologie, Cologne
  - HELIOS Klinikum Erfurt, Erfurt
  - Universitatsklinikum Essen, Essen
  - Universitätsmedizin Göttingen, Göttingen
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinik Heidelberg, Heidelberg
  - UKSH Kiel, Kiel
  - Universitätsklinikum Leipzig, Leipzig
  - UKSH Universitatsklinikum Schleswig-Holstein, Lübeck
  - Universitatsklinikum Mainz, Mainz
  - Klinikum der Ludwigs-Maximilians-Universität München, München
  - Fachklinik Hornheide, Münster
  - Harzklinikum Dorothea Christiane Erxleben GmbH, Standort Quedlinburg, Quedlinburg
  - Universitätsklinikum Regensburg, Regensburg
  - Zentrum für Dermatoonkologie, Universitäts-Hautklinik Tübingen, Tübingen
  - Universitätsklinikum Würzburg, Würzburg
- Greece (2):
  - Laiko General Hospital Athen, Athens
  - Metropolitan Hospital, Pireaus
- Hungary (2):
  - Orszagos Onkologiai Intezet, Budapest
  - University of Szeged Szent-Györgyi Albert Clinical Center, Szeged
- Israel (4):
  - Rambam Health Care Campus, Haifa
  - Sharett Institute - Hadassah Hebrew University Medical Center, Jerusalem
  - Rabin MC, Petah Tikva
  - Ella Institute - Sheba Medical Center, Ramat Gan
- Italy (10):
  - Istituto Tumori ?Giovanni Paolo II?, Oncologia, Bari, Apulia
  - IRCCS Istituto Nazionale Tumori Fondazione Pascale, Napoli, Campania
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola, Meldola, Emilia-Romagna
  - A.O. Universitaria S. Maria Della Misericordia Di Udine, Udine, Friuli Venezia Giulia
  - IFO - Istituto Regina Elena, Rome, Lazio
  - IRCCS Istituto Nazionale Per La Ricerca Sul Cancro (IST), Genoa, Liguria
  - Irccs Istituto Nazionale Dei Tumori (Int), Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO), Milan, Lombardy
  - Fondazione Del Piemonte Per L'oncologia Ircc Di Candiolo, Candiolo, Piedmont
  - A.O.U. Senese Policlinico Santa Maria Alle Scotte, Siena, Tuscany
- Erasmus Mc - Daniel Den Hoed Kliniek, Rotterdam, Netherlands
- New Zealand (3):
  - Wellington Hospital, Newtown, Wellington
  - Mid Central DHB, Palmerston North
  - Tauranga Hospital, Clinical Trials Unit, Tauranga
- Poland (6):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Narodowy Inst.Onkol.im.Sk?odowskiej-Curie Pa?stw.Inst.Badawczy Kraków, Krakow
  - COZL Oddzial Onkologii Klinicznej z pododdzialem Chemioterapii Dziennej, Lublin
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Późna
  - Narodowy Instytut Onkologii im. Marii Sk?odowskiej-Curie - Pa?stwowy Instytut Badawczy, Warsaw
  - Dolno?l?skie Centrum Onkologii, Pulmonologii i Hematologii, Wroclaw
- Portugal (2):
  - IPO de Lisboa, Lisbon
  - IPO do Porto, Porto
- Russia (3):
  - Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast
  - FSBSI "Russian Oncological Scientific Center n.a. N.N. Blokhin", Moscow, Moscow Oblast
  - FBI "Scientific Research Institute of Oncology n. a. N. N. Petrov", Saint Petersburg, Sankt-Peterburg
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (9):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic i Provincial, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Macarena, Seville
  - Fundacion Instituto Valenciano de Oncologia (IVO), Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (8):
  - Bristol Haematology and Oncology centre, Bristol
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Ipswich Hospital, Ipswich
  - St James Uni Hospital, Leeds
  - Guys and St Thomas NHS Foundation Trust, Guys Hospital, London
  - Freeman Hospital, New Castle Upon Tyne
  - Singleton Hospital, Swansea
  - Royal Cornwall Hospital, Truro

REFERENCES:
- [Derived] Li SN, Wan X, Peng LB, Li YM, Li JH. Cost-effectiveness of immune checkpoint inhibition and targeted treatment in combination as adjuvant treatment of patient with BRAF-mutant advanced melanoma. BMC Health Serv Res. 2023 Jan 18;23(1):49. doi: 10.1186/s12913-023-09058-7. PMID 36653848
- [Derived] Ascierto PA, Stroyakovskiy D, Gogas H, Robert C, Lewis K, Protsenko S, Pereira RP, Eigentler T, Rutkowski P, Demidov L, Zhukova N, Schachter J, Yan Y, Caro I, Hertig C, Xue C, Kusters L, McArthur GA, Gutzmer R. Overall survival with first-line atezolizumab in combination with vemurafenib and cobimetinib in BRAFV600 mutation-positive advanced melanoma (IMspire150): second interim analysis of a multicentre, randomised, phase 3 study. Lancet Oncol. 2023 Jan;24(1):33-44. doi: 10.1016/S1470-2045(22)00687-8. Epub 2022 Nov 29. PMID 36460017
- [Derived] Robert C, Lewis KD, Gutzmer R, Stroyakovskiy D, Gogas H, Protsenko S, Pereira RP, Eigentler T, Rutkowski P, Demidov L, Caro I, Forbes H, Shah K, Yan Y, Li H, McArthur GA, Ascierto PA. Biomarkers of treatment benefit with atezolizumab plus vemurafenib plus cobimetinib in BRAFV600 mutation-positive melanoma. Ann Oncol. 2022 May;33(5):544-555. doi: 10.1016/j.annonc.2022.01.076. Epub 2022 Feb 4. PMID 35131452
- [Derived] de Azevedo SJ, de Melo AC, Roberts L, Caro I, Xue C, Wainstein A. First-line atezolizumab monotherapy in patients with advanced BRAFV600 wild-type melanoma. Pigment Cell Melanoma Res. 2021 Sep;34(5):973-977. doi: 10.1111/pcmr.12960. Epub 2021 Feb 15. PMID 33476492
- [Derived] Gutzmer R, Stroyakovskiy D, Gogas H, Robert C, Lewis K, Protsenko S, Pereira RP, Eigentler T, Rutkowski P, Demidov L, Manikhas GM, Yan Y, Huang KC, Uyei A, McNally V, McArthur GA, Ascierto PA. Atezolizumab, vemurafenib, and cobimetinib as first-line treatment for unresectable advanced BRAFV600 mutation-positive melanoma (IMspire150): primary analysis of the randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2020 Jun 13;395(10240):1835-1844. doi: 10.1016/S0140-6736(20)30934-X. PMID 32534646

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 514 participants with B-Raf proto-oncogene serine/threonine kinase (BRAF) V600 mutation positive metastatic or unresectable locally advanced melanoma took part in the study. The study had 2 periods: 28-day run-in period & a triple combination period.
  The study was closed early by the sponsor due to the low likelihood of OS achieving statistical significance at final analysis & slower-than-anticipated OS event accumulation. Hence, the study was considered to be completed.
Pre-assignment Details: Participants received either Placebo + Cobimetinib + Vemurafenib (Pbo+Cobi+Vem) or Atezolizumab + Cobimetinib + Vemurafenib (Atezo+Cobi+Vem). 26 participants were included in pbo+cobi+vem arm for safety analysis (22 in atezo+cobi+vem arm stopped run-in treatment & received no atezo & 4 in atezo+cobi+vem arm completed the run-in treatment but did not receive atezo). During the study, 2 participants in pbo+cobi+vem arm received atezo & were included in the atezo+cobi+vem arm for safety analysis.
Groups:
- Run-in - Pbo + Cobi + Vem: Participants received vemurafenib, 960 milligrams (mg) (four, 240 mg tablets), orally (PO), twice a day (BID) along with cobimetinib, 60 mg (three, 20 mg tablets) PO, once a day (QD) on Days 1 to 21 only followed by vemurafenib 960 mg (four, 240 mg tablets), PO, BID on Days 22 to 28 during the 28 day run-in period.
- Run-in - Atezo + Cobi + Vem: Participants received vemurafenib, 960 mg (four, 240 mg tablets) PO, BID along with cobimetinib 60 mg (three, 20 mg tablets) PO, QD on Days 1 to 21 only followed by vemurafenib 720 mg (three, 240 mg tablets) PO, BID and vemurafenib matching placebo, PO, BID on Days 22 to 28 during the 28 day run-in period.
- Triple Combination: Pbo + Cobi + Vem: After the 28-day run-in, participants received atezolizumab matching placebo as IV infusion on Days 1 and 15, cobimetinib, 60 mg (three, 20 mg tablets) PO, QD, on Days 1 to 21 and vemurafenib 960 mg (four, 240 mg tablets) PO, BID on Days 1 to 28. Study treatment was continued until investigator determined disease progression (PD), death, unacceptable toxicity, withdrawal of consent, or pregnancy, whichever occurred first.
- Triple Combination: Atezo + Cobi + Vem: After the 28-day run-in period, participants received atezolizumab 840 mg as IV infusion on Days 1 and 15, cobimetinib, 60 mg (three, 20 mg tablets) PO, QD, on Days 1 to 21, vemurafenib 720 mg (three, 240 mg tablets) PO BID on Days 1 to 28, and vemurafenib placebo (1 tablet) PO BID on Days 1 to 28. Study treatment was continued until investigator determined PD, death, unacceptable toxicity, withdrawal of consent, or pregnancy, whichever occurred first.
Period: Run-in Period
Arm/Group | Run-in - Pbo + Cobi + Vem | Run-in - Atezo + Cobi + Vem | Triple Combination: Pbo + Cobi + Vem | Triple Combination: Atezo + Cobi + Vem
Started | 258 | 256 | 0 | 0
Completed | 234 | 234 | 0 | 0
Not Completed | 24 | 22 | 0 | 0
Not completed — Death | 12 | 10 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Reason Not Specified | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Not completed — Study Ended by Sponsor | 5 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 9 | 0 | 0
Period: Triple Combination Period
Arm/Group | Run-in - Pbo + Cobi + Vem | Run-in - Atezo + Cobi + Vem | Triple Combination: Pbo + Cobi + Vem | Triple Combination: Atezo + Cobi + Vem
Started | 0 | 0 | 231 | 230
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 231 | 230
Not completed — Death | 0 | 0 | 150 | 127
Not completed — Lost to Follow-up | 0 | 0 | 6 | 8
Not completed — Reason Not Specified | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 1
Not completed — Study Ended by Sponsor | 0 | 0 | 61 | 77
Not completed — Withdrawal by Subject | 0 | 0 | 13 | 16

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all randomized participants, whether or not study treatment was received.
Groups:
- Arm A: Pbo + Cobi + Vem: Participants received vemurafenib, 960 mg (four, 240 mg tablets), PO, BID along with cobimetinib, 60 mg (three, 20 mg tablets) PO, QD on Days 1 to 21 only followed by vemurafenib 960 mg (four, 240 mg tablets), PO, BID on Days 22 to 28 during the 28 day run-in period. During triple combination period (Cycle 1 onwards), participants received atezolizumab matching placebo as IV infusion on Days 1 and 15, cobimetinib, 60 mg (three, 20 mg tablets) PO, QD, on Days 1 to 21 and vemurafenib 960 mg (four, 240 mg tablets) PO, BID on Days 1 to 28. Study treatment was continued until investigator determined PD, death, unacceptable toxicity, withdrawal of consent, or pregnancy, whichever occurred first.
- Arm B: Atezo + Cobi + Vem: Participants received vemurafenib, 960 mg (four, 240 mg tablets) PO, BID along with cobimetinib 60 mg (three, 20 mg tablets) PO, QD on Days 1 to 21 only followed by vemurafenib 720 mg (three, 240 mg tablets) PO, BID and vemurafenib matching placebo, PO, BID on Days 22 to 28 during the 28 day run-in period. During triple combination period (Cycle 1 onwards), participants received atezolizumab 840 mg as IV infusion on Days 1 and 15, cobimetinib, 60 mg (three, 20 mg tablets) PO, QD, on Days 1 to 21, vemurafenib 720 mg (three, 240 mg tablets) PO BID on Days 1 to 28, and vemurafenib placebo (1 tablet) PO BID on Days 1 to 28. Study treatment was continued until investigator determined PD, death, unacceptable toxicity, withdrawal of consent, or pregnancy, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Arm A: Pbo + Cobi + Vem | Arm B: Atezo + Cobi + Vem | Total
Number analyzed (Participants) | 258 | 256 | 514
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 199 | 195 | 394
  >=65 years | 59 | 61 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (14.1) | 54.0 (14.2) | 53.6 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 106 | 215
  Male | 149 | 150 | 299
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 27 | 47
  Not Hispanic or Latino | 225 | 223 | 448
  Unknown or Not Reported | 13 | 6 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 4 | 7 | 11
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 1 | 1
  White | 246 | 243 | 489
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS), as Determined by Investigator Using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: PFS was defined as the time from randomization to the first occurrence of PD, as determined by the investigator according to RECIST v1.1, or death from any cause, whichever occurred first. PD was defined as at least a 20% increase in the sum of diameters (SOD) of target lesions, taking as reference smallest sum on study, including baseline. In addition to the relative increase of 20%, the SOD must also demonstrate an absolute increase of at least 5 millimeters (mm).
Time Frame: Baseline up to PD or death due to any cause, whichever occurred first (up to approximately 33 months)
Population: ITT population included all randomized participants, whether or not study treatment was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Pbo + Cobi + Vem | Arm B: Atezo + Cobi + Vem
Number analyzed (Participants) | 258 | 256
months | 10.6 [9.3 to 12.7] | 15.1 [11.4 to 18.4]
Statistical Analysis 1: Comparison: Arm A: Pbo + Cobi + Vem vs Arm B: Atezo + Cobi + Vem; Test type: Superiority; p = 0.0224, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.64 to 0.97] — Stratified Hazard Ratio

2. Secondary Outcome: PFS as Determined by Independent Review Committee (IRC) Using RECIST v1.1
Description: PFS was defined as the time from randomization to the first occurrence of disease progression, as determined by the IRC according to RECIST v1.1, or death from any cause, whichever occurred first. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference smallest sum on study, including baseline. In addition to the relative increase of 20%, the SOD must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Baseline up to PD or death due to any cause, whichever occurred first (up to approximately 33 months)
Population: ITT population included all randomized participants, whether or not study treatment was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Pbo + Cobi + Vem | Arm B: Atezo + Cobi + Vem
Number analyzed (Participants) | 258 | 256
months | 12.3 [10.8 to 14.7] | 16.1 [11.3 to 18.5]
Statistical Analysis 1: Comparison: Arm A: Pbo + Cobi + Vem vs Arm B: Atezo + Cobi + Vem; Test type: Superiority; p = 0.1607, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.67 to 1.07] — Stratified Hazard Ratio

3. Secondary Outcome: Percentage of Participants With Objective Response (OR), as Determined by Investigator Using RECIST V1.1
Description: OR rate was defined as percentage of participants with partial response (PR) or complete response (CR) on 2 consecutive occasions ≥ 4 weeks apart as determined by the investigator using RECIST v.1.1. CR was defined as the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD.
Time Frame: Baseline up to PD or death due to any cause, whichever occurred first (up to approximately 56 months)
Population: ITT population included all randomized participants, whether or not study treatment was received. Only participants with measurable disease at baseline were analyzed for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Pbo + Cobi + Vem | Arm B: Atezo + Cobi + Vem
Number analyzed (Participants) | 246 | 255
percentage of participants | 65.0 | 66.7
Statistical Analysis 1: Comparison: Arm A: Pbo + Cobi + Vem vs Arm B: Atezo + Cobi + Vem; Test type: Superiority; p = 0.6997, Cochran-Mantel-Haenszel; Difference in response rate = 1.63, 95% CI 2-sided [-6.90 to 10.15]

4. Secondary Outcome: Duration of Response (DOR), as Determined by Investigator Using RECIST v1.1
Description: DOR was defined as the time from the first occurrence of a documented OR to PD, as determined by the investigator according to RECIST v1.1, or death from any cause, whichever occurred first. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference smallest sum on study, including baseline. In addition to the relative increase of 20%, the SOD must also demonstrate an absolute increase of at least 5 mm. CR was defined as the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD.
Time Frame: Baseline up to PD or death due to any cause, whichever occurred first (up to approximately 56 months)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Pbo + Cobi + Vem | Arm B: Atezo + Cobi + Vem
Number analyzed (Participants) | 246 | 255
months | 12.6 [10.5 to 16.7] | 21.0 [16.6 to 32.2]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death from any cause.
Time Frame: Baseline up to death due to any cause (up to approximately 85 months)
Population: ITT population included all randomized participants, whether or not study treatment was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Pbo + Cobi + Vem | Arm B: Atezo + Cobi + Vem
Number analyzed (Participants) | 258 | 256
months | 25.8 [22.0 to 34.6] | 39.0 [29.9 to 55.3]
Statistical Analysis 1: Comparison: Arm A: Pbo + Cobi + Vem vs Arm B: Atezo + Cobi + Vem; Test type: Superiority; p = 0.1191, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.67 to 1.05]

6. Secondary Outcome: Percentage of Participants Who Have Survived at 2 Years
Description: Percentage of participants with OS which was defined as the time from randomization to death from any cause. The Kaplan-Meier approach was used to estimate 2-year landmark survival rate. The 95% CI of landmark survival rate was calculated using the standard error derived from Greenwood's formula.
Time Frame: 2 years
Population: ITT population included all randomized participants, whether or not study treatment was received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Pbo + Cobi + Vem | Arm B: Atezo + Cobi + Vem
Number analyzed (Participants) | 258 | 256
percentage of participants | 53.31 [47.00 to 59.62] | 61.50 [55.31 to 67.70]
Statistical Analysis 1: Comparison: Arm A: Pbo + Cobi + Vem vs Arm B: Atezo + Cobi + Vem; Test type: Superiority; p = 0.0693, Z-test; Difference in Event Free Rate = 8.20, 95% CI 2-sided [-0.65 to 17.04]

7. Secondary Outcome: Time to Deterioration in Global Health Status (GHS) Determined Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Scale Score
Description: Time to deterioration in GHS/health related quality of life (HRQoL) was defined as the time from randomization to first observed ≥ 10-point decrease in EORTC QLQ-C30 linearly transformed GHS/HRQoL scale score that is sustained for two consecutive assessments or followed by death while the participant is on treatment. EORTC QLQ-C30 consists of 30 questions that assess five aspects of participant functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, pain), GHS/QoL, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The GHS/QoL are scored on a 7-point scale (1=Very Poor to 7=Excellent). The obtained scores are linearly transformed to a score range of 0-100, where higher scores indicate a higher response level and better QoL.
Time Frame: Baseline up to PD or death due to any cause, whichever occurred first (up to approximately 33 months)
Population: ITT population included all randomized participants, whether or not study treatment was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Pbo + Cobi + Vem | Arm B: Atezo + Cobi + Vem
Number analyzed (Participants) | 258 | 256
months | NA [15.0 to NA] — Median and upper limit of 95% CI were not estimable due to an insufficient number of participants with event. | 14.4 [9.2 to NA] — Upper limit of 95% CI was not estimable due to an insufficient number of participants with event.

8. Secondary Outcome: Time to Deterioration in Physical Functioning (PF) Determined Using EORTC QLQ-C30 Scale Score
Description: Time to deterioration in PF = time from randomization to first observed ≥ 10-point decrease in EORTC QLQ-C30 linearly transformed PF scale score that is sustained for two consecutive assessments or followed by death while the participant is on treatment. EORTC QLQ-C30 consists of 30 questions that assess 5 aspects of participant functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, pain), GHS/QoL, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). PF scale has 5 questions about participant's PF and daily activities (strenuous activities, long walks, short walks, bed/chair rest & needing help with eating, dressing, washing themselves, or using the toilet). PF are scored on a 4-point scale (1=Not at All to 4=Very Much). The obtained scores are linearly transformed to a score range of 0-100, where higher scores indicate a higher response level, functioning/support.
Time Frame: Baseline up to PD or death due to any cause, whichever occurred first (up to approximately 33 months)
Population: ITT population included all randomized participants, whether or not study treatment was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Pbo + Cobi + Vem | Arm B: Atezo + Cobi + Vem
Number analyzed (Participants) | 258 | 256
months | 22.4 [15.7 to NA] — Upper limit of 95% CI was not estimable due to an insufficient number of participants with event. | 17.5 [11.7 to NA] — Upper limit of 95% CI was not estimable due to an insufficient number of participants with event.

9. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant when administered a pharmaceutical product regardless of the causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with the use of an investigational product, whether or not considered related to the investigational product. A SAE is any significant hazard, contraindication, side effect that is fatal or life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is medically significant or requires intervention to prevent one or other of the outcomes listed above. All AEs were reported until 30 days and SAEs until 90 days after the final dose of study treatment or until initiation of subsequent anti-cancer therapy, whichever occurred first.
Time Frame: Up to approximately 85 months
Population: Safety population included all participants who received any amount of any atezolizumab, cobimetinib, or vemurafenib. 26 were included in the placebo+cobi+vem arm for safety evaluation (22 participants in atezo+cobi+vem arm stopped run-in treatment & didn't received atezo & 4 in atezo+cobi+vem arm completed the run-in treatment but did not receive atezo). During the study, 2 participants in placebo+cobi+vem arm received atezo & were considered in the atezo+cobi+vem arm for safety analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Pbo + Cobi + Vem | Arm B: Atezo + Cobi + Vem
Number analyzed (Participants) | 279 | 232
percentage of participants
  AEs | 99.6 | 100
  SAEs | 43.0 | 50.9

10. Secondary Outcome: Serum Concentration of Atezolizumab
Time Frame: Pre-infusion Day 1 of Cycles 1-4; 30 minutes post-infusion Day 1 of Cycles 1 and 4; at Atezolizumab discontinuation (up to approximately 33 months) (1 Cycle = 28 days)
Population: Pharmacokinetic (PK)-evaluable population included all participants who have received any dose of atezolizumab and for whom at least one evaluable PK sample was collected. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per milliliters (ug/mL)
Arm/Group | Arm B: Atezo + Cobi + Vem
Number analyzed (Participants) | 223
micrograms per milliliters (ug/mL)
  Cycle 1 Day 1/30 Min Postdose: number analyzed (Participants) | 187
  Cycle 1 Day 1/30 Min Postdose | 281 (111)
  Cycle 2 Day 1/Predose: number analyzed (Participants) | 186
  Cycle 2 Day 1/Predose | 102 (47.4)
  Cycle 3 Day 1/Predose: number analyzed (Participants) | 171
  Cycle 3 Day 1/Predose | 149 (61.9)
  Cycle 4 Day 1/Predose: number analyzed (Participants) | 159
  Cycle 4 Day 1/Predose | 181 (75.5)
  Cycle 4 Day 1/30 Min Postdose: number analyzed (Participants) | 144
  Cycle 4 Day 1/30 Min Postdose | 431 (158)
  Study Drugs Discontinuation Visit: number analyzed (Participants) | 101
  Study Drugs Discontinuation Visit | 122 (97.7)

11. Secondary Outcome: Plasma Concentration of Cobimetinib Dose: 20/40 mg
Time Frame: Pre-dose (0 hour) and 3 to 6 hours post dose on Day 15 of Cycles 1 and 4 (1 Cycle = 28 days)
Population: The Cobi PK-evaluable population included all participants who received any dose of cobimetinib 20/40 mg and for whom at least one evaluable PK sample was collected. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Arm A: Pbo + Cobi + Vem | Arm B: Atezo + Cobi + Vem
Number analyzed (Participants) | 218 | 208
mg
  Cycle 1 Day 15/Predose: number analyzed (Participants) | 32 | 29
  Cycle 1 Day 15/Predose | 79.9 (72.2) | 144 (101)
  Cycle 1 Day 15/3-6 Hr Postdose: number analyzed (Participants) | 32 | 26
  Cycle 1 Day 15/3-6 Hr Postdose | 167 (116) | 216 (145)
  Cycle 4 Day 15/Predose: number analyzed (Participants) | 43 | 49
  Cycle 4 Day 15/Predose | 108 (97.5) | 92.3 (79.5)
  Cycle 4 Day 15/3-6 Hr Postdose: number analyzed (Participants) | 45 | 47
  Cycle 4 Day 15/3-6 Hr Postdose | 167 (126) | 171 (140)

12. Secondary Outcome: Plasma Concentration of Cobimetinib Dose: 60 mg
Time Frame: Pre-dose (0 hour) and 3 to 6 hours post dose on Day 15 of Cycles 1 and 4 (1 Cycle = 28 days)
Population: The Cobi PK-evaluable population included all participants who received any dose of Cobimetinib 60 mg and for whom at least one evaluable PK sample was collected. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Arm A: Pbo + Cobi + Vem | Arm B: Atezo + Cobi + Vem
Number analyzed (Participants) | 218 | 208
mg
  Cycle 1 Day 15/Predose: number analyzed (Participants) | 170 | 148
  Cycle 1 Day 15/Predose | 169 (171) | 216 (188)
  Cycle 1 Day 15/3-6 Hr Postdose: number analyzed (Participants) | 171 | 140
  Cycle 1 Day 15/3-6 Hr Postdose | 278 (206) | 375 (243)
  Cycle 4 Day 15/Predose: number analyzed (Participants) | 123 | 112
  Cycle 4 Day 15/Predose | 150 (113) | 151 (120)
  Cycle 4 Day 15/3-6 Hr Postdose: number analyzed (Participants) | 120 | 109
  Cycle 4 Day 15/3-6 Hr Postdose | 240 (195) | 256 (197)

13. Secondary Outcome: Plasma Concentration of Vemurafenib
Time Frame: Pre-dose (0 hour) and 3 to 6 hours post dose on Day 15 of Cycles 1 and 4 (1 Cycle = 28 days)
Population: The Vem PK-evaluable population included all participants who received any dose of vemurafenib and for whom at least one evaluable PK sample was collected. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Arm A: Pbo + Cobi + Vem | Arm B: Atezo + Cobi + Vem
Number analyzed (Participants) | 218 | 209
μg/mL
  Cycle 1 Day 15/ predose: number analyzed (Participants) | 199 | 179
  Cycle 1 Day 15/ predose | 38.9 (100) | 27.0 (102)
  Cycle 1 Day 15/ 3-6 hr: number analyzed (Participants) | 205 | 168
  Cycle 1 Day 15/ 3-6 hr | 41.3 (57.7) | 28.0 (88.6)
  Cycle 4 Day 15/ predose: number analyzed (Participants) | 168 | 158
  Cycle 4 Day 15/ predose | 39.2 (105) | 24.7 (202)
  Cycle 4 Day 15/ 3-6 hr postdose: number analyzed (Participants) | 168 | 154
  Cycle 4 Day 15/ 3-6 hr postdose | 42.3 (59.4) | 26.5 (135)

14. Secondary Outcome: Percentage of Participants Positive for Anti-drug Antibodies (ADA) to Atezolizumab
Description: Presence of ADAs against atezolizumab during the study relative to the presence of ADAs at baseline. The percentage of ADA-positive participants after drug administration were determined for participants exposed to atezolizumab. For determining post-baseline incidence, participants were considered to be ADA-positive if they were ADA-negative or had missing data at baseline but developed an ADA response following study drug exposure, or if they were ADA-positive at baseline and the titer of 1 or more post-baseline samples was at least 0.60 titer units (t.u.) greater than the baseline titer result.
Time Frame: Pre-infusion Day 1 of Cycles 1-4 (1 Cycle=28 days); at Atezolizumab discontinuation (approximately up to 33 months)
Population: The ADA-evaluable population included participants who received at least one dose of atezolizumab and had ≥ 1 post-baseline ADA result. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Arm B: Atezo + Cobi + Vem
Number analyzed (Participants) | 218
percentage of participants
  Baseline evaluable participants: number analyzed (Participants) | 208
  Baseline evaluable participants | 1.4
  Post-baseline evaluable participants | 13.3

ADVERSE EVENTS:
Time Frame: Run-in Period: 28 days Triple Combination Period: From the first dose of study treatment in the Triple Combination Period (Day 29) up to approximately 85 months
Description: 26 participants were included in the placebo+cobi+vem arm for safety evaluation (22 participants in atezo+cobi+vem arm stopped run-in treatment & received no atezo & 4 in atezo+cobi+vem arm completed the run-in treatment but did not receive atezo). During the study, 2 participants in placebo+cobi+vem arm received atezo & were considered in the atezo+cobi+vem arm for safety analysis. Of the 26 participants who were considered in placebo for safety, 10 died and hence are shown in the placebo arm.
Groups:
- Run-in - Pbo + Cobi + Vem: Participants received vemurafenib, 960 mg (four, 240 mg tablets), PO, BID along with cobimetinib, 60 mg (three, 20 mg tablets) PO, QD on Days 1 to 21 only followed by vemurafenib 960 mg (four, 240 mg tablets), PO, BID on Days 22 to 28 during the 28 day run-in period.
- Triple Combination: Pbo + Cobi + Vem: After the 28-day run-in, participants received atezolizumab matching placebo as IV infusion on Days 1 and 15, cobimetinib, 60 mg (three, 20 mg tablets) PO, QD, on Days 1 to 21 and vemurafenib 960 mg (four, 240 mg tablets) PO, BID on Days 1 to 28. Study treatment was continued until investigator determined PD, death, unacceptable toxicity, withdrawal of consent, or pregnancy, whichever occurred first.
Arm/Group | Run-in - Atezo + Cobi + Vem | Run-in - Pbo + Cobi + Vem | Triple Combination: Pbo + Cobi + Vem | Triple Combination: Atezo + Cobi + Vem
All-Cause Mortality (participants affected / at risk) | 0/232 | 25/279 | 149/279 | 128/232
Serious Adverse Events (participants affected / at risk) | 21/232 | 50/279 | 81/279 | 109/232
Other Adverse Events (participants affected / at risk) | 208/232 | 262/279 | 222/279 | 226/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in - Atezo + Cobi + Vem (N=232) | Run-in - Pbo + Cobi + Vem (N=279) | Triple Combination: Pbo + Cobi + Vem (N=279) | Triple Combination: Atezo + Cobi + Vem (N=232)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Central serous chorioretinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Detachment of retinal pigment epithelium (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Maculopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal artery embolism (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Autoimmune colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 7 (7) | 6 (7) | 13 (18)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Autoimmune cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Hepatitis fulminant (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Bacterial prostatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bartholin's abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 2 (2) | 2 (3) | 4 (4)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Large intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 8 (11)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serratia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 5 (6) | 2 (2) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain dislocation syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalitis autoimmune (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated encephalitis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 6 (6)
Nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian rupture (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in - Atezo + Cobi + Vem (N=232) | Run-in - Pbo + Cobi + Vem (N=279) | Triple Combination: Pbo + Cobi + Vem (N=279) | Triple Combination: Atezo + Cobi + Vem (N=232)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 9 (11) | 37 (62) | 44 (78)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 13 (19) | 17 (47)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 28 (31) | 48 (62)
Hypothyroidism (Endocrine disorders) | 2 (2) | 3 (3) | 23 (24) | 46 (67)
Central serous chorioretinopathy (Eye disorders) | 9 (9) | 19 (19) | 27 (34) | 25 (33)
Dry eye (Eye disorders) | 0 (0) | 2 (2) | 2 (2) | 14 (15)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 12 (14) | 13 (18)
Vision blurred (Eye disorders) | 3 (3) | 8 (9) | 12 (17) | 12 (15)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 9 (11) | 22 (39) | 28 (44)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 11 (11) | 21 (29) | 20 (23)
Constipation (Gastrointestinal disorders) | 9 (10) | 21 (21) | 16 (24) | 30 (36)
Diarrhoea (Gastrointestinal disorders) | 78 (90) | 113 (131) | 85 (186) | 74 (196)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 2 (2) | 10 (10) | 16 (17)
Dyspepsia (Gastrointestinal disorders) | 8 (8) | 5 (5) | 16 (23) | 14 (17)
Nausea (Gastrointestinal disorders) | 37 (38) | 41 (41) | 64 (96) | 55 (97)
Stomatitis (Gastrointestinal disorders) | 12 (15) | 6 (6) | 11 (15) | 15 (30)
Vomiting (Gastrointestinal disorders) | 16 (18) | 31 (31) | 45 (72) | 45 (63)
Asthenia (General disorders) | 11 (12) | 19 (22) | 36 (68) | 50 (101)
Chills (General disorders) | 8 (9) | 13 (13) | 11 (19) | 18 (20)
Fatigue (General disorders) | 34 (35) | 38 (41) | 56 (84) | 50 (74)
Influenza like illness (General disorders) | 2 (3) | 4 (4) | 12 (14) | 19 (24)
Mucosal inflammation (General disorders) | 7 (7) | 5 (5) | 12 (16) | 12 (25)
Oedema peripheral (General disorders) | 9 (10) | 13 (14) | 27 (36) | 45 (59)
Pain (General disorders) | 1 (1) | 1 (1) | 8 (8) | 13 (14)
Pyrexia (General disorders) | 46 (55) | 48 (54) | 58 (120) | 93 (203)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 5 (7) | 13 (16)
Conjunctivitis (Infections and infestations) | 0 (0) | 3 (3) | 13 (14) | 19 (21)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 12 (19) | 12 (13)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 10 (13) | 18 (27)
Nasopharyngitis (Infections and infestations) | 4 (4) | 3 (3) | 27 (41) | 21 (41)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 4 (4) | 22 (23) | 23 (28)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3) | 10 (17) | 21 (45)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 18 (24) | 24 (31)
Sunburn (Injury, poisoning and procedural complications) | 12 (14) | 10 (10) | 26 (50) | 21 (47)
Alanine aminotransferase increased (Investigations) | 14 (14) | 24 (25) | 52 (69) | 73 (127)
Amylase increased (Investigations) | 9 (9) | 17 (20) | 40 (72) | 46 (91)
Aspartate aminotransferase increased (Investigations) | 14 (14) | 20 (22) | 42 (61) | 66 (133)
Blood alkaline phosphatase increased (Investigations) | 13 (15) | 19 (20) | 33 (46) | 33 (70)
Blood bilirubin increased (Investigations) | 6 (6) | 8 (8) | 11 (18) | 24 (75)
Blood creatine phosphokinase increased (Investigations) | 48 (52) | 67 (74) | 96 (308) | 108 (328)
Blood creatinine increased (Investigations) | 17 (17) | 17 (17) | 35 (62) | 42 (119)
Blood lactate dehydrogenase increased (Investigations) | 4 (4) | 5 (5) | 9 (15) | 19 (32)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 11 (12) | 13 (16)
Ejection fraction decreased (Investigations) | 1 (1) | 2 (2) | 6 (6) | 13 (14)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 5 (5) | 16 (21) | 15 (20)
Lipase increased (Investigations) | 21 (25) | 20 (27) | 75 (200) | 77 (184)
Weight decreased (Investigations) | 2 (2) | 7 (7) | 8 (12) | 13 (13)
Decreased appetite (Metabolism and nutrition disorders) | 12 (12) | 19 (20) | 25 (38) | 25 (29)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 7 (7) | 11 (23) | 18 (37)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (6) | 4 (5) | 12 (17) | 12 (14)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (5) | 3 (3) | 15 (27) | 14 (49)
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 (34) | 42 (48) | 70 (134) | 84 (193)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 18 (20) | 26 (32)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 8 (9) | 14 (18)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (18) | 12 (14) | 42 (62) | 52 (80)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (9) | 8 (8) | 25 (38) | 29 (51)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 15 (22) | 7 (9)
Dizziness (Nervous system disorders) | 4 (4) | 4 (4) | 12 (13) | 15 (16)
Dysgeusia (Nervous system disorders) | 7 (7) | 5 (5) | 6 (6) | 15 (17)
Headache (Nervous system disorders) | 11 (11) | 16 (16) | 45 (71) | 55 (95)
Insomnia (Psychiatric disorders) | 4 (4) | 5 (5) | 17 (19) | 13 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (8) | 26 (32) | 35 (63)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 18 (19) | 18 (28)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (5) | 10 (12) | 24 (26)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 13 (18) | 29 (36)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 14 (22) | 4 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 25 (27) | 24 (24)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 12 (13) | 28 (28) | 23 (34) | 29 (43)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6) | 7 (7) | 21 (24) | 28 (30)
Erythema (Skin and subcutaneous tissue disorders) | 10 (10) | 15 (17) | 33 (51) | 36 (42)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 8 (13) | 12 (13)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 16 (16) | 40 (42) | 45 (66) | 40 (63)
Pruritus (Skin and subcutaneous tissue disorders) | 24 (28) | 18 (19) | 34 (66) | 53 (104)
Rash (Skin and subcutaneous tissue disorders) | 62 (67) | 81 (96) | 63 (106) | 71 (121)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 31 (34) | 44 (51) | 10 (11) | 19 (28)
Hypertension (Vascular disorders) | 11 (11) | 21 (21) | 39 (52) | 36 (45)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/72/NCT02908672/Prot_001.pdf
  • Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT02908672/SAP_002.pdf